CLINICAL TRIAL: NCT04293900
Title: Prospective Observational Study of Diet, Physical Activity and Body Composition Changes During R-CHOP Treatment for NHL
Brief Title: Diet, Physical Activity and Body Composition Changes During R-CHOP
Acronym: R-CHOP-OS
Status: Withdrawn | Type: Observational
Why Stopped: Study never started due to COVID pandemic and lack of study funding.
Sponsor: George Washington University (Other)
Responsible Party: Principal Investigator, Kimberly Robien, Associate Professor, George Washington University
Other Study IDs: 180373
Record Dates: First submitted 2020-02-18; First posted 2020-03-03 (Actual); Last update posted 2020-10-06 (Actual); Status verified 2020-10

CONDITIONS: Non-Hodgkin Lymphoma; DLBCL; Diffuse Large B Cell Lymphoma
Keywords: diet; physical activity; body composition; bisphenol; phthalate; gut microbiome
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Lymphoma, Large B-Cell, Diffuse; Motor Activity | interventions — Hand Strength

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — urine, fecal samples (optional component of the study)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Study cohort: 24-hour dietary recall, hand grip strength, accelerometer, International Physical Activity Questionnaire (IPAQ), Patient-reported outcomes survey (NCI-PRO-CTCAE), Pittsburgh Sleep Quality Index (PSQI), Functional Assessment of Cancer Treatment - Lymphoma (FACT-lym), urine sample (optional), fecal sample (optional)
  Interventions: Other: 24-hour dietary recall; Other: Hand grip strength; Other: International Physical Activity Questionnaire; Other: Patient-reported outcomes survey; Other: Pittsburgh Sleep Quality Index; Other: Functional Assessment of Cancer Treatment - Lymphoma; Other: urine sample (optional); Other: fecal sample (optional)

INTERVENTIONS:
Other: 24-hour dietary recall — Dietary intake assessment conducted by a Registered Dietitian Nutritionist. This assessment will occur prior to starting R-CHOP chemotherapy, during the clinic visits for each round of R-CHOP chemotherapy, and again at the end of the scheduled course of R-CHOP chemotherapy.
Other: Hand grip strength — Measurement of grip strength using a hand dynamometer. This will test occur prior to starting R-CHOP chemotherapy, during the clinic visits for each round of R-CHOP chemotherapy, and again at the end of the scheduled course of R-CHOP chemotherapy.
Other: International Physical Activity Questionnaire — Survey about physical activity over the previous 7 days. This survey will be administered prior to starting R-CHOP chemotherapy, during the clinic visits for each round of R-CHOP chemotherapy, and again at the end of the scheduled course of R-CHOP chemotherapy.
  Other Names: IPAQ
Other: Patient-reported outcomes survey — Survey about symptoms and side effects experienced during cancer treatment. This will be administered prior to starting R-CHOP chemotherapy, during the clinic visits for each round of R-CHOP chemotherapy, and again at the end of the scheduled course of R-CHOP chemotherapy.
  Other Names: NCI-PRO-CTCAE
Other: Pittsburgh Sleep Quality Index — Survey about sleep habits and quality over the past month. This will be administered prior to starting R-CHOP chemotherapy, during the clinic visits for each round of R-CHOP chemotherapy, and again at the end of the scheduled course of R-CHOP chemotherapy.
  Other Names: PSQI
Other: Functional Assessment of Cancer Treatment - Lymphoma — Survey about quality of life for people with a diagnosis of lymphoma. This will be administered prior to starting R-CHOP chemotherapy, during the clinic visits for each round of R-CHOP chemotherapy, and again at the end of the scheduled course of R-CHOP chemotherapy.
  Other Names: FACT-lym
Other: urine sample (optional) — Collect three urine samples either in the clinic or at home. This specimen collection will occur prior to starting R-CHOP chemotherapy, after the third round of R-CHOP chemotherapy, and again at the end of the scheduled course of R-CHOP chemotherapy.
Other: fecal sample (optional) — Collect a fecal sample either in the clinic or at home. This sample collection will occur prior to starting R-CHOP chemotherapy, after the third round of R-CHOP chemotherapy, and again at the end of the scheduled course of R-CHOP chemotherapy.

SUMMARY:
In this pilot study, observational data will be collected to describe the usual trajectory of changes in dietary intake, ability to be physically active, body composition, environmental exposures, and the gut microbiome over the course of R-CHOP treatment for non-Hodgkin lymphoma (NHL).

DETAILED DESCRIPTION:
Rituximab plus cyclophosphamide, doxorubicin, vincristine, and prednisone (R-CHOP) is the "gold standard" first-line treatment for patients with non-Hodgkin lymphoma, yet it is estimated that R-CHOP is not curative for 30- 50% of patients. Preliminary studies suggests that modifiable lifestyle factors such as body composition, exposure to endocrine disrupting chemicals, and changes in the gut microbiome may contribute to variation in R-CHOP treatment response. If true, it could be possible to modify these factors in an effort to improve treatment outcomes, however more detailed information is needed to confirm these preliminary findings and test whether lifestyle modification can improve outcomes.

In this observational study, data will be collected on dietary intake, ability to be physically active, body composition, environmental exposure to endocrine disrupting chemicals and changes in the gut microbiome over the course of R-CHOP for NHL. The study will provide more detailed information on the usual trajectory of these lifestyle factors during R-CHOP treatment than has previously been collected, especially how these factors co-vary over time. The study findings are expected to inform future intervention studies aimed at improving R-CHOP treatment outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of one of the non-Hodgkin lymphomas
* Scheduled to receive R-CHOP at the George Washington University Cancer Center

Exclusion Criteria:

* Diagnosis of cancer other than one of the non-Hodgkin lymphomas
* Patients who are scheduled to receive their R-CHOP somewhere other than the George Washington University Cancer Center
* Patients who are not competent to provide informed consent to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients being treated at the George Washington University for non-Hodgkin lymphoma who are scheduled to receive R-CHOP chemotherapy
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2021-01 (Estimated); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Change in lean body mass (LBM) from baseline to end of R-CHOP chemotherapy | baseline and post-R-CHOP chemotherapy (18 weeks)
  change in kilograms of lean body mass as measured from staging CT-scans from pre- to post-R-CHOP chemotherapy.

SECONDARY OUTCOMES:
Change in adipose tissue volume from baseline to end of R-CHOP chemotherapy | baseline and post-R-CHOP chemotherapy (18 weeks)
  change in adipose tissue volume (cm^3) as measured from staging CT-scans from pre- to post-R-CHOP chemotherapy.
Change in dietary energy from baseline to end of R-CHOP chemotherapy | baseline, each chemotherapy visit (3, 6, 9, 12, and 15 weeks), and post-R-CHOP chemotherapy (18 weeks)
  Change in total energy intake (kcal/day) from pre- to post-R-CHOP chemotherapy.
Change in dietary protein intake from baseline to end of R-CHOP chemotherapy | baseline, each chemotherapy visit (3, 6, 9, 12, and 15 weeks), and post-R-CHOP chemotherapy (18 weeks)
  Change in dietary protein intake (g/day) from pre- to post-R-CHOP chemotherapy measured by diet history.
Change in physical activity level from baseline to end of R-CHOP chemotherapy | baseline, each chemotherapy visit (3, 6, 9, 12, and 15 weeks), and post-R-CHOP chemotherapy (18 weeks)
  Change in daily metabolic equivalents (MET) of physical activity as measured by accelerometer from pre- to post-R-CHOP chemotherapy.
Change in urinary bisphenol levels | baseline, after the third chemotherapy visit (9 weeks), and post-R-CHOP chemotherapy (18 weeks)
  percent of change in urinary bisphenol levels (ng/mL) as measured by liquid chromotography-tandem mass spectrometry from pre- to post-R-CHOP chemotherapy
Change in urinary phthalate levels | baseline, after the third chemotherapy visit (9 weeks), and post-R-CHOP chemotherapy (18 weeks)
  percent of change in urinary phthalate levels (ng/ML) as measured by liquid chromotography-tandem mass spectrometry from pre- to post-R-CHOP chemotherapy
Change in gut microbiome composition | baseline, after the third chemotherapy visit (9 weeks), and post-R-CHOP chemotherapy (18 weeks)
  Change in species and type of gut microbiota from pre- to post-R-CHOP chemotherapy

CONTACTS AND LOCATIONS:
Overall Officials: Kim Robien, PhD, RD, Principal Investigator — Milken Institute School of Public Health, George Washington University
Locations (1):
- Milken Institute School of Public Health, George Washington University, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: No
Will not share data until study is complete and all data deidentified